CLINICAL TRIAL: NCT05583786
Title: Intracoronary ECG ST-segment Shift Remission Time During Reactive Coronary Hyperemia, τ-icECG: a New Method for Assessing Hemodynamic Stenosis Severity
Brief Title: Intracoronary ECG ST-segment Shift Remission Time During Reactive Coronary Hyperemia
Acronym: τ-icECG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00522
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Chronic Coronary Syndrome
Keywords: Intracoronary electrocardiogram; icECG; Reactive-hyperemia; Balloon occlusion; Fractional flow ratio; FFR
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tracing intracoronary electrocardiogram — icECG ST-segment shift remission time (τ-icECG) tracing during reactive-hyperemia, obtained immediately after a 1-minute upstream coronary artery balloon occlusion.

SUMMARY:
This study evaluates a new diagnostic approach based on intracoronary electrocardiogram (icECG) ST-segment shift remission time, denoted as τ-icECG (τ=tau, i.e., the remission half-time fitted by an exponential function to the disappearing ST-segment shift), to be used for PCI guidance.

DETAILED DESCRIPTION:
Cardiovascular disease is the major cause of death globally, accounting for 17.9 million deaths per year in 2019. Aside from the acute coronary syndrome, where percutaneous coronary intervention (PCI) has been shown to improve outcome, the number of patients with chronic coronary syndrome (CCS) is also increasing. PCI of hemodynamically relevant stenotic lesions causing myocardial ischemia is the standard treatment in these patients. Effective revascularization, as recommended by the European Society of Cardiology (ESC) guidelines, requires to differentiate between hemodynamically relevant and non-significant stenotic coronary lesions.

Currently, coronary stenosis assessment is performed by structural visual angiographic assessment or by coronary pressure measurements up- and downstream of the lesion. The latter is recommended by the ESC and is based on its prognostic value derived from large randomized clinical trials. Given temporary paralysis of the coronary microcirculation by a hyperemia-inducing substance such as adenosine (ADO), pressure is, in theory, directly related to coronary flow. Therefore, the pressure drop during hyperemia across a coronary stenosis, i.e., fractional flow reserve (FFR) provides an estimate of its restrictive effect on flow. However, this method depends on expensive pressure sensor angioplasty guidewires, and on hyperemia-inducing substances, such as ADO. Hence, pharmacologic limitations such as atrioventricular conduction defects and asthma and other potential adverse events (e.g. arrhythmias) aside from costs are major drawbacks of pressure-derived FFR. In order to avoid potential drug-induced side effects and achieve maximal hyperemia, the study group performs reactive hyperemia FFR measurements induced by a proximal, 1-minute coronary artery balloon occlusion. This method has been documented non-inferior in its ability to detect relevant coronary stenosis compared to adenosine-induced FFR.

The present project aims at validating a novel, potentially more harmless, faster and less costly diagnostic approach for measuring hemodynamic coronary stenosis severity.

The commonly obtained surface lead electrocardiogram (ECG) is limited in detecting short-lasting or minor myocardial ischemia. In comparison, intracoronary ECG (icECG) is more time- and space-sensitive in detecting myocardial ischemia, the latter being due to its close vicinity to the myocardial region of interest. It can be easily obtained by attaching an alligator clamp to a coronary guidewire.

Based on the sensitivity of the icECG, several clinical trials have assessed the value of icECG to guide PCI, and rated it useful to predict post-procedural myocardial injury.

The investigators research group performed a trial to determine the diagnostic accuracy of icECG ST-segment shift during pharmacologic inotropic stress in assessing functional coronary lesion severity versus structural stenosis severity as obtained by quantitative coronary angiography in % diameter narrowing (%S by QCA), and versus other functional hemodynamic indices (FFR, instantaneous wave-free ratio (iFR)). IcECG ST-segment shift showed a significant correlation with all established parameters.

Evaluation of icECG required the development of a specific software algorithm, which robustly determines quantitative icECG ST-segment shift in every single heartbeat. The validation analysis of the algorithm took place in an offline setting and demonstrated an excellent correlation as compared to the results of ECG experts (r2 = 0.932; p<0.001).

The development of this fully autonomous icECG analyzing algorithm was set up on an existing ECG software, denoted as "EsoLive", developed at the Institute for Medical Engineering and Medical Informatics, University of Applied Sciences and Arts Northwestern Switzerland. In short, the algorithm starts with a baseline wander extraction method related to Kalman filtering, then sets the initial points for an "edge", i.e., J-point, before, it processes in a similar way the isoelectric line level. Quantitative time as well as voltage measurements of those two points allow the calculation of the icECG ST-segment shift for each single QRS complex.

This study evaluates a new diagnostic approach based on icECG ST-segment shift remission time, denoted as τ-icECG (τ=tau, i.e., the remission half-time fitted by an exponential function to the disappearing ST-segment shift), to be used for PCI guidance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary syndrome
* Chronic stable 1-3 vessel coronary artery disease
* Coronary stenotic lesion of any diameter narrowing
* Age > 18 years
* Referred for elective coronary angiography to the investigators institution
* Written informed consent to participate in the study

Exclusion Criteria:

* Acute coronary syndrome
* Unstable cardiopulmonary condition
* Severe aortic valve stenosis
* Acute congestive heart failure NYHA (New York Heart Association) III-IV
* ECG bundle branch blocks, non-sinus rhythm or paced rhythm
* Coronary anatomy unsuitable for coronary measurements
* Severe pulmonary, renal or hepatic disease
* Women of childbearing age (≤50years and ≤12months after the last menstruation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic coronary syndrome electively referred to the investigators department for coronary angiography.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
icECG ST-segment shift remission time (τ-icECG) | once after a 1-minute coronary ballon occlusion
  The primary study objective is to test reactive hyperemia τ-icECG as obtained immediately after a 1-minute upstream coronary artery balloon occlusion as a new method to determine the hemodynamic significance of a coronary artery stenosis. As primary reference method, reactive hyperemia FFR (cut-off 0.80) is employed.

SECONDARY OUTCOMES:
Quantitative percent diameter narrowing (secondary reference) (%S) | once after a 1-minute coronary ballon occlusion
  The secondary study objective is to test reactive hyperemia τ-icECG against the structural reference of a coronary artery stenosis, %S, and to compare the accuracy of τ-icECG against reactive hyperemia FFR, and instantaneous wave-free ratio (iFR).
Reactive hyperemia FFR (primary reference) | once after a 1-minute coronary ballon occlusion
  The secondary study objective is to compare the accuracy of τ-icECG against reactive hyperemia FFR.
Instantaneous wave-free ratio (iFR) | once before a 1-minute coronary ballon occlusion
  The secondary study objective is to compare the accuracy of τ-icECG against iFR.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, Prof, Principal Investigator — Inselspital
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta SR, Cannon CP, Fox KA, Wallentin L, Boden WE, Spacek R, Widimsky P, McCullough PA, Hunt D, Braunwald E, Yusuf S. Routine vs selective invasive strategies in patients with acute coronary syndromes: a collaborative meta-analysis of randomized trials. JAMA. 2005 Jun 15;293(23):2908-17. doi: 10.1001/jama.293.23.2908. PMID 15956636
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Stegehuis VE, Wijntjens GW, Piek JJ, van de Hoef TP. Fractional Flow Reserve or Coronary Flow Reserve for the Assessment of Myocardial Perfusion : Implications of FFR as an Imperfect Reference Standard for Myocardial Ischemia. Curr Cardiol Rep. 2018 Jul 26;20(9):77. doi: 10.1007/s11886-018-1017-4. PMID 30046914
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] Piccolo R, Niglio T, Di Gioia G, D'Anna C, De Rosa R, Strisciuglio T, Trimarco B, Piscione F, Galasso G. Adenosine-induced torsade de pointes complicating a fractional flow reserve measurement in a right coronary artery intermediate stenosis. Cardiovasc Revasc Med. 2013 Mar-Apr;14(2):118-20. doi: 10.1016/j.carrev.2012.12.010. Epub 2013 Feb 19. PMID 23433828
- [Background] Stoller M, Seiler C. Reactive myocardial hyperaemia for functional assessment of coronary stenosis severity. EuroIntervention. 2017 Jun 2;13(2):e201-e209. doi: 10.4244/EIJ-D-16-00579. PMID 27993753
- [Background] Friedman PL, Shook TL, Kirshenbaum JM, Selwyn AP, Ganz P. Value of the intracoronary electrocardiogram to monitor myocardial ischemia during percutaneous transluminal coronary angioplasty. Circulation. 1986 Aug;74(2):330-9. doi: 10.1161/01.cir.74.2.330. PMID 2942314
- [Background] Pande AK, Meier B, Urban P, Moles V, Dorsaz PA, Favre J. Intracoronary electrocardiogram during coronary angioplasty. Am Heart J. 1992 Aug;124(2):337-41. doi: 10.1016/0002-8703(92)90595-m. PMID 1636577
- [Background] Hishikari K, Yonetsu T, Lee T, Koura K, Murai T, Iwai T, Takagi T, Isobe M, Iesaka Y, Kakuta T. Intracoronary electrocardiogram ST-segment elevation in patients with non-ST-segment elevation myocardial infarction and its association with culprit lesion location and myocardial injury. EuroIntervention. 2014 May;10(1):105-12. doi: 10.4244/EIJV10I1A17. PMID 24048173
- [Background] Balian V, Galli M, Marcassa C, Cecchin G, Child M, Barlocco F, Petrucci E, Filippini G, Michi R, Onofri M. Intracoronary ST-segment shift soon after elective percutaneous coronary intervention accurately predicts periprocedural myocardial injury. Circulation. 2006 Oct 31;114(18):1948-54. doi: 10.1161/CIRCULATIONAHA.106.620476. Epub 2006 Oct 23. PMID 17060382
- [Background] Bigler MR, Stoller M, Praz F, Siontis GCM, Grossenbacher R, Tschannen C, Seiler C. Functional assessment of myocardial ischaemia by intracoronary ECG. Open Heart. 2021 Jan;8(1):e001447. doi: 10.1136/openhrt-2020-001447. PMID 33462106